CLINICAL TRIAL: NCT03780166
Title: A Phase 2 Dose-Escalation Study of the Safety and Tolerability of INCB050465 in Participants With Pemphigus Vulgaris
Brief Title: A Study of the Safety and Tolerability of INCB050465 in Pemphigus Vulgaris
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to insufficient interest in study participation due to recent approval in this rare condition.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-208; Parsaclisib (Other: Incyte Corporation)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Pemphigus Vulgaris
Keywords: Pemphigus vulgaris; phosphatidylinositol 3-kinase delta; immunoglobulin G autoantibodies
MeSH Terms: conditions — Pemphigus | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Parsaclisib (Experimental)
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib administered orally once daily at the cohort-specified dose level.
  Other Names: INCB050465

SUMMARY:
The purpose of this study is to assess the safety and tolerability of parsaclisib in participants with mild to moderate pemphigus vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Clinically documented and confirmed diagnosis of pemphigus vulgaris: minimum of 6 months of pemphigus vulgaris diagnosis; positive for anti-desmoglein (DSG)1 or DSG3; Pemphigus Disease Area Index score of 8 to 45 points; active skin, scalp, or mucosal lesions.
* Disease progression after treatment with standard therapies that are known to confer clinical benefit, or intolerant to treatment; there is no limit to the number of prior treatment regimens.
* Willingness to avoid pregnancy or fathering children.
* If required, willing to receive Pneumocystis jirovecii pneumonia prophylaxis during the study period.

Exclusion Criteria:

* Pregnant or breast-feeding female.
* Participants with pemphigus vulgaris who are treatment-naive.
* Use of protocol-specified medications within defined periods before baseline.
* Evidence or history of clinically significant infection or protocol-defined medical conditions
* Laboratory values outside the protocol-defined range at screening.
* Known or suspected allergy to parsaclisib or any component of the study drug.
* Known history of clinically significant drug or alcohol abuse in the last year before baseline.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to 20 weeks
  Any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.

SECONDARY OUTCOMES:
Cmax of Parsaclisib | Up to 6 weeks
  Maximum observed concentration.
tmax of Parsaclisib | Up to 6 weeks
  Time to maximum concentration.
Cmin of Parsaclisib | Up to 6 weeks
  Minimum observed concentration over the dose interval.
AUC0-t of Parsaclisib | Up to 6 weeks
  Area under the concentration-time curve from time = 0 to the last measurable concentration at time = t.
CL/F of Parsaclisib | Up to 6 weeks
  Apparent oral dose clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation

IPD SHARING:
Plan to Share IPD: No